CLINICAL TRIAL: NCT04424264
Title: The Effect of Rifampicin on the Pharmacokinetics of Intracellular Tenofovir-diphosphate and Tenofovir When Coadministered With Tenofovir Alafenamide Fumarate During the Maintenance Phase of Tuberculosis Treatment in TB/HIV-1 Coinfected Participants
Acronym: EpiTAF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Professor Francois Venter (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor-Investigator, Professor Francois Venter, Divisional Director of Ezintsha, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WRHI061
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: HIV-1-infection; Tuberculosis
Keywords: Rifampicin, RIF/INH; Tenofovir alafenamide fumarate (TAF); Pharmacokinetics; Intracellular tenofovir-diphosphate
MeSH Terms: conditions — Tuberculosis | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tenofovir Alafenamide (Experimental): TAF 25 mg once-daily administered with RIF/INH 600*/300mg
  Interventions: Drug: Phase 1: Tenofovir disoproxil fumarate/Emtricitabine/Efavirenz coadministered with Rifampicin/Isoniazid; Drug: Phase 2: Tenofovir alafenamide/Lamivudine/Efavirenz coadministered with Rifampicin/Isoniazid; Drug: Phase 3: Tenofovir disoproxil fumarate/Emtricitabine/Efavirenz

INTERVENTIONS:
Drug: Phase 1: Tenofovir disoproxil fumarate/Emtricitabine/Efavirenz coadministered with Rifampicin/Isoniazid — TDF/FTC/EFV 300/200/600 mg once daily plus RIF/INH 600*/300 mg daily from screening until enrolment (days -15 to 0)
  Other Names: Atripla; Rifinah
Drug: Phase 2: Tenofovir alafenamide/Lamivudine/Efavirenz coadministered with Rifampicin/Isoniazid — TAF 25 mg + 3TC 300 mg + EFV 600 mg once daily plus RIF/INH 600/*300 mg daily (days 1 to ≤ 56)
  Other Names: HepBest; Stocrin
Drug: Phase 3: Tenofovir disoproxil fumarate/Emtricitabine/Efavirenz — TDF/FTC/EFV 300/200/600 mg once daily. RIF/INH 600mg <70kg, 750mg >70kg
  Other Names: Atripla; Rifinah

SUMMARY:
This is a pharmacokinetic study investigating the effect of rifampicin on the pharmacokinetics of intracellular tenofovir-diphosphate and plasma tenofovir when coadministered with tenofovir alafenamide fumarate during the maintenance phase of tuberculosis treatment in TB/HIV-1 coinfected participants (EpiTAF)

DETAILED DESCRIPTION:
This is an open-label, sequential, single centre pharmacokinetic (PK) study investigating the effect of rifampicin on the pharmacokinetics of intracellular tenofovir-diphosphate and plasma tenofovir when coadministered with tenofovir alafenamide fumarate during the maintenance phase of tuberculosis treatment in TB/HIV-1 coinfected participants (EpiTAF).

An open-label, sequential, pharmacokinetic (PK) drug-drug interaction study will be conducted in medically stable virologically suppressed HIV-1 infected adults coinfected with TB, who are in the maintenance phase of their TB treatment. After intensive PK evaluation of IC TFV-DP and pTFV, participants will be switched from their standard-of-care tenofovir disoproxil fumarate (TDF)/FTC/EFV regimen, to TAF + 3TC + EFV at the start of the study treatment period. After 28 days each participant will have intensive PK evaluation of IC TFV-DP and pTFV on TAF + 3TC + EFV with rifampicin (RIF). After the second intensive PK assessment is completed, participants will be switched back to TDF/FTC/EFV, with a final intensive PK evaluation of IC TFV-DP and pTFV 8 days after completion of TB treatment, at the final study visit. Eighteen volunteers will be enrolled for a target of 13 participants completing the study.

The study includes screening and enrolment visits, 1 visit on day 28 and an end of study visit 28 days after the end of TB treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years old) male or female
2. HIV-1 infected on TDF/FTC/EFV with HIV RNA < 50 copies/mL in the last three months
3. On TB treatment in the maintenance phase (RIF/INH) with at least one month of TB treatment needed for completion
4. Women of childbearing potential must not be pregnant or breastfeeding, with a negative pregnancy test at screening
5. Women must be postmenopausal, surgically sterile or practicing an effective birth control method (established before and maintained throughout the trial). Women who are not sexually active must agree to use an effective birth control method if they become heterosexually active during the trial
6. Understand the purpose of and procedures required for the study and having confirmed they are willing to participate in the study by signing the informed consent document.

Exclusion Criteria:

1. Weight < 40 kg
2. Estimated creatinine clearance < 50 mL/min
3. Any active clinically significant or life-threatening disease (e.g. acute infections, pancreatitis, hepatitis, cardiac dysfunction), medical or psychiatric condition, or findings during screening, that in the investigator's opinion would compromise the safety of the participant or the study outcome, or their ability to comply with the study procedures
4. Chronic medical requirement for any drugs that are known to affect the PK of the study drugs
5. Active drug/alcohol abuser
6. History of allergy or hypersensivity to any of the study drugs
7. Currently enrolled in an investigational drug study or has participated in an investigational drug study within the 4 weeks before screening
8. Unable to comply with study protocol and study protocol restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
IC TFV-DP concentrations during coadministration of TAF or TDF with RIF/INH in TB/HIV-1 coinfected participants | 56 days
  Intracellular and plasma TFV-DP concentrations measured during coadministration of TAF or TDF with RIF/INH

SECONDARY OUTCOMES:
Maintenance of irological suppression (HIV-1 RNA < 50 copies/mL) | At screening, day 28, completion of TB and EOS visits
  Assessment of maintenance of virological suppression (HIV-1 RNA < 50 copies/mL) while on TAF/RIF
Comparison plasma concentrations of TAF with TDF | 56 days
  Assessment to compare the plasma concentrations of tenofovir of TAF with TDF during coadministration of RIF/INH in TB/HIV-1 coinfected participants
Comparison of IC TFV-DP concentrations of TDF | 56 days
  4. To compare the IC TFV-DP concentrations of TDF with and without coadministration with RIF/INH in TB/HIV-1 coinfected participants

CONTACTS AND LOCATIONS:
Overall Officials: Simiso Sokhela, MBBCh, Principal Investigator — Ezintsha, a subdivision of Wits Reproductive Health and HIV Institute (Wits RHI)
Locations (2):
- South Africa (2):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Wits RHI Yeoville Clinic, Johannesburg, Gauteng